CLINICAL TRIAL: NCT01399502
Title: Promotion of Self-help Strategies for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orygen (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Melbourne (Other); Sidney Myer Fund (Unknown)
Responsible Party: Principal Investigator, Amy Morgan, PhD candidate, Orygen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0931313
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Depressive Disorder; Depression
Keywords: Depression; Self Care
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-help advice (Active Comparator): Each email will contain a self-help strategy for coping with depressive symptoms. The email will contain information about why the strategy will be effective, tips for implementing the strategy and overcoming barriers, and how to set a goal to implement the strategy. Strategies are based on previous research published by the trial co-ordinators.
  Interventions: Behavioral: Mood Memo emails
- Depression information (Placebo Comparator): Each email will contain different information about depression, such as symptoms, risk factors, prevalence.
  Interventions: Behavioral: Mood Memo emails

INTERVENTIONS:
Behavioral: Mood Memo emails — Participants will receive 12 emails over 6 weeks.

SUMMARY:
The purpose of this study is to investigate the effectiveness of health promotion emails for depression. It is hypothesised that emails containing self-help advice will improve depression symptoms more than emails containing information about depression.

DETAILED DESCRIPTION:
Depression symptoms are commonly experienced and disrupt day-to-day life. Increasing depression literacy and the use of effective self-help methods could improve depression across the community. The internet is an ideal promotional medium for health messages, because it is often used to search for information about mental health issues, and health messages can be widely disseminated at little cost. An email campaign could be a low-cost approach to improving self-help behavior and knowledge about depression in adults with depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Access to the internet at least once per week
* Resident of Australia, New Zealand, Canada, Ireland, United Kingdom, USA

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1736 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Depression symptom score on PHQ-9 at post-intervention | 6-weeks post baseline
Depression symptom score on PHQ-9 at 6-month follow-up | 6-months post end-of-intervention

SECONDARY OUTCOMES:
Psychological distress on K10 at post-intervention | 6-weeks post baseline
Psychological functioning on Work and Social Adjustment Scale at post-intervention | 6-weeks post baseline
Psychological functioning on Work and Social Adjustment Scale at 6-month follow-up | 6-months post end-of-intervention
Psychological distress on K10 at 6-month follow-up | 6-months post end-of-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Jorm, PhD, DSc, Principal Investigator — Orygen Youth Health Research Centre, The University of Melbourne; Andrew J Mackinnon, PhD, Principal Investigator — Orygen Youth Health Research Centre, The University of Melbourne
Locations (1):
- Orygen Youth Health Research Centre, Parkville, Victoria, Australia

REFERENCES:
- [Derived] Morgan AJ, Jorm AF, Mackinnon AJ. Self-Help for Depression via E-mail: A Randomised Controlled Trial of Effects on Depression and Self-Help Behaviour. PLoS One. 2013 Jun 21;8(6):e66537. doi: 10.1371/journal.pone.0066537. Print 2013. PMID 23805231